CLINICAL TRIAL: NCT02645032
Title: A Randomized, Observer-Blinded, Phase I Study to Assess the Safety and Immunogenicity of Vi-DT Conjugate Vaccine Compared to Vi-Polysaccharide (Typhim Vi®, Sanofi Pasteur) Typhoid Vaccine in Healthy Filipino Adults and Children
Brief Title: Safety and Immunogenicity of a Vi-DT Typhoid Conjugate Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI T001
Record Dates: First submitted 2015-12-22; First posted 2016-01-01 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2018-02

CONDITIONS: Typhoid
Keywords: Typhoid conjugate vaccine; Vi-DT; Safety; Immunogenicuty
MeSH Terms: conditions — Typhoid Fever | interventions — Vi polysaccharide vaccine, typhoid; vaxigrip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Laboratory personnel who analyzes immunogenicity at sponsor is also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Two doses of Vi-DT (typhoid conjugate vaccine) will be administrated intramuscularly 4 weeks apart (Day 0 and Day 28).
  Interventions: Biological: Vi-DT
- Comparator group (Active Comparator): Biological/Vaccine:
  One dose of Typhim Vi® will be administrated intramuscularly at 1st dose (Day 0).
  One dose of VAXIGRIP® will be administrated intramuscularly at 2nd dose (Day 28).
  Interventions: Biological: Typhim Vi®; Biological: VAXIGRIP®

INTERVENTIONS:
Biological: Vi-DT — Manufacturer: SK Chemicals Co., Ltd. Ingredient: Purified Vi-polysaccharide conjugated to diphtheria toxoid Dose: 0.5 mL/Vial
  Other Names: Vi-DT typhoid conjugate vaccine
  Arms: Test group
Biological: Typhim Vi® — Manufacturer: Sanofi Pasteur Ingredient: Purified Vi-polysaccharide Appearance: colourless liquid Dose: 0.5mL/vial
  Arms: Comparator group
Biological: VAXIGRIP® — Dose: Single injection, participants 6-35 months of age will receive 0.25 ml (half a dose), participants 36 months of age and older will receive 0.5ml (full dose)
  *Participants less than 9 years of age, who have not been vaccinated for flu before, will receive a second dose of flu-vaccine after the last follow-up visit of last participant in their age cohort.
  Arms: Comparator group

SUMMARY:
This is a Phase I, Randomized, observer-blinded, age de-escalating study.

The study objectives are:

1. To evaluate the safety of 25 μg of Vi-DT typhoid conjugate vaccine administered at 0 and 4 weeks.
2. To assess the immunogenicity of 25 μg of Vi-DT typhoid conjugate vaccine administered at 0 and 4 weeks.
3. To compare the safety and immunogenicity of Vi-DT and Vi-Polysaccharide typhoid vaccines.

DETAILED DESCRIPTION:
This study will be carried out in healthy adults and children at a single site. Subjects will be stratified according to age.

The study procedure is as follows:

Visit 1 (day-1 to -7): Screen participants by medical history, physical examination and lab investigations. Collect blood for safety and immunogenicity assessments.

Visit 2 (day 0): Enroll, randomize and administer first dose of vaccine to eligible participants

Visit 3 (day 3): Assess participant safety by medical history and physical examination

Visit 4 (day 7): Record solicited adverse reaction 7 days post vaccination, and collect blood for safety lab assessments.

Visit 5 (day 28): Assess participant safety, collect blood for immunogenicity assessments, and administer second vaccine dose

Visit 6 (day 31): Participants safety will be assessed by medical history and physical examination

Visit 7 (day 35): Record solicited adverse reaction 7 days post second vaccination.

Visit 8 (day 56): Collect blood for immunogenicity assessments, assess participant safety, and fill in study completion form in the absence of any safety concern.

This study is observer-blind: vaccine administrator and vaccine safety evaluator will be two distinct persons to avoid bias of safety assessment. Trial staff other than the vaccine administrator.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female individual 2-45 years of age
2. Participants/Parents who have voluntarily given informed consent and/or assent.
3. Participants/Parents willing to commit complying with the study procedures of the investigator and available for the entire duration of study

Exclusion Criteria:

1. Participants concomitantly enrolled or scheduled to be enrolled in another trial
2. Acute illness, in particular infectious diseases or fever (axillary temperature > 38°C), with in three days prior to enrollment and vaccination.
3. Known history of allergy to vaccines or other medications
4. Known history of allergy to egg, chiken protein, neomycin and formaldehyde.
5. History of uncontrolled coagulopathy or blood disorders
6. Known history of immune function disorders including immunodeficiency diseases, or chronic use of systemic steroids (> 20 mg/day prednisone equivalent for periods exceeding 10 days), cytotoxic or other immunosuppressive drugs
7. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the participant and interfere with the assessment of the trial objectives
8. Pregnancy & Lactation (female adults)
9. Female with child-bearing potential during the study period. i.e., sexually active and not practicing effective acceptable contraceptive method
10. Individuals who have previously received any vaccines against typhoid fever
11. Individuals already immunized with any licensed vaccine within 4 weeks prior to enrolment/vaccination (day 0) and expected to receive other licensed vaccines within 60 days following the first dose (day 0), except for tetanus toxoid vaccine
12. Individuals who have a previously ascertained or suspected disease caused by S. typhi.
13. Individuals who have had household contact with/and or intimate exposure to an individual with laboratory-confirmed S. typhi
14. History of alcohol or substance abuse
15. Subject planning to move from the study area before the end of study period

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Safety endpoints for solicited adverse events (reactogenicity) and serious adverse events | 4 weeks post first and second vaccination
  Proportion of participants with local and systemic solicited adverse events (reactogenicity) and Proportion of participant with Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Proportion of participants with sero-conversion | 4 weeks post first and second injections of Vi-DT and one injection of Vipolysaccharide
  Defined as a four-fold rise in anti-Vi antibody titers compared to baseline measured by anti-Vi IgG ELISA and Serum Bactericidal Assay
Geometric Mean Titers (GMT) | 4 weeks post first and second vaccination
  Measurement of the Geometric Mean Titers (GMT) following 4 weeks post first and second injections of Vi-DT and one injection of Vi-polysaccharide vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario Capeding, MD, Principal Investigator — Research Institution for Tropical Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capeding MR, Teshome S, Saluja T, Syed KA, Kim DR, Park JY, Yang JS, Kim YH, Park J, Jo SK, Chon Y, Kothari S, Yang SY, Ham DS, Ryu JH, Hwang HS, Mun JH, Lynch JA, Kim JH, Kim H, Excler JL, Sahastrabuddhe S. Safety and immunogenicity of a Vi-DT typhoid conjugate vaccine: Phase I trial in Healthy Filipino adults and children. Vaccine. 2018 Jun 18;36(26):3794-3801. doi: 10.1016/j.vaccine.2018.05.038. PMID 29776750
- See also: Final Result — https://doi.org/10.1016/j.vaccine.2018.05.038